CLINICAL TRIAL: NCT05200377
Title: Magnetic Resonance Imaging in Cerebral Small Vessel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Department of Radiology, Chinese PLA General Hospital
Other Study IDs: ChinaPLAGH-Radiology
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Small Vessel Diseases; MRI
Keywords: Cerebral small vessel diseases; Cognitive impairments; Lesion burden; MRI
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cerebral small vessel disease group: Patients with clinically and radiologically evidenced cerebral small vessel disease. Patients are grouped by severity of cerebral small vessel disease assessed by comprehensive MRI findings.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Patients recruited will receive Magnetic resonance imaging.

SUMMARY:
Cerebral small vessel disease (cSVD) accounts for 20% of ischemic strokes and is the most common cause of vascular cognitive impairment. Early identification of cSVD is critical for early intervention and improve clinical outcomes. Magnetic resonance imaging (MRI) may represent as a sensitive and robust tool to detect early changes in brain subtle structures and functions. The study is to investigate the comprehensive evaluation of brain structures and vascular functions by using advanced MRI technologies in early diagnosis and management of cSVD.

DETAILED DESCRIPTION:
Cerebral small vessel disease (cSVD) accounts for 20% of ischemic strokes and is the most common cause of vascular cognitive impairment. Early identification of cSVD is critical for early intervention and improve clinical outcomes. Magnetic resonance imaging (MRI) is sensitive to change in white matter structure and subtle vascular function alternation which correlates with cognition impairments in cSVD. MRI manifestation may also represent as useful surrogate marker. Development of advanced MRI technologies promotes their invaluable application in brain and vascular qualitative and quantitative assessment. The study is to investigate the comprehensive evaluation of brain structures and vascular functions by using advanced MRI technologies in early diagnosis and management of cSVD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of cerebral small vessel disease or MRI evidence of lacunar infarcts and white matter hyperintensity
* No disability (modified Rankin's scale < 2)
* No dementia (MMSE > 24 and absence of dependence in daily activities)
* Able and willing to consent

Exclusion Criteria:

* Contraindications to MRI
* Standard MRI of bad quality due to movement artefacts
* Pregnant
* Unable to tolerate MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinically or radiologically evidenced cerebral small vessel disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression in total cerebral small vessel disease burden | 1 year
  Total cSVD burden assessed by MRI

SECONDARY OUTCOMES:
Progression in congnitive impairments | 1 years
  Global Z-score by cognitive domain
Recurrent ischemic events | 1 year
  Recurrent ischemic stroke, TIA and vascular death
Modified Rankin Scale | 90 days and 1 year after qualifying event
  Disability assessed by modified Rankin Scale (mRS). The scores, ranging from 0 (no symptoms) to 6 (death), were recorded by phone call or outpatient consultation. A favorable outcome was defined as mRS score 0-2, unfavorable outcome was defined as mRS score > 2.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wardlaw JM, Smith C, Dichgans M. Small vessel disease: mechanisms and clinical implications. Lancet Neurol. 2019 Jul;18(7):684-696. doi: 10.1016/S1474-4422(19)30079-1. Epub 2019 May 13. PMID 31097385
- [Derived] Duan C, Bian X, Cheng K, Lyu J, Xiong Y, Xiao S, Wang X, Duan Q, Li C, Huang J, Hu J, Wang ZJ, Zhou X, Lou X. Synthesized 7T MPRAGE From 3T MPRAGE Using Generative Adversarial Network and Validation in Clinical Brain Imaging: A Feasibility Study. J Magn Reson Imaging. 2024 May;59(5):1620-1629. doi: 10.1002/jmri.28944. Epub 2023 Aug 9. PMID 37559435